CLINICAL TRIAL: NCT03980886
Title: Characteristics and Inflammatory Markers in Children with Eosinophilic Esophagitis (EoE)
Acronym: EoE
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Seema Aceves, Professor, Pediatrics and Medicine, University of California, San Diego
Other Study IDs: 181690; 2R56AI092135 (NIH); 2R01DK114457 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-06-10 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Esophageal biopsies and/or cells derived from biopsies and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Single center observational and specimen banking study for children with eosinophilic esophagitis EoE to gauge natural history and inflammatory markers

DETAILED DESCRIPTION:
Participants with a diagnosis of EoE are recruited from Rady Children's Hospital Eosinophilic Gastrointestinal Disorders (EGID) during routine clinic and/or endoscopy visits.

Medical information including clinical symptoms, endoscopy, histopathology, medical and surgical history, lab and imaging findings, are entered into a UCSD database at each clinic or endoscopy visit. Blood and biopsy specimens are procured and utilized for analysis of inflammatory molecules and for isolation of structural cells. This protocol continues our clinical database and sample collection in children with EoE. The database provides a cohort of EoE patients for studies of natural history, therapeutic response, and disease progression. In a relatively new disease of increasing incidence, these studies will provide information on disease progression and the clinical characteristics of patients who have varying disease phenotypes as well as the associations between clinical phenotypes, molecular changes, and disease course. The procurement and storage of tissue, cells, and serum samples provides a repository for studies of EoE-related molecules and peripheral markers in clinically phenotyped patients. In addition, the study of these esophageal cells will provide an in vitro model system for assessing the molecular mechanisms of disease pathogenesis in EoE.

ELIGIBILITY:
Inclusion Criteria:

* Have a known EoE diagnosis
* Complain of dysphagia, vomiting, or abdominal pain, especially if recalcitrant to acid blocking therapy (but does not have to be recalcitrant to acid blocking medications)
* Present with food impaction
* Present with esophageal stricture
* Have characteristic endoscopic findings of EoE of pallor, linear furrows, lichenification, white plaques, or concentric rings

Exclusion Criteria:

* None

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The majority of patients who are diagnosed with EoE or suspected EoE at RCHSD/UCSD
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2028-12-17 (Estimated); Study Completion 2028-12-17 (Estimated)

PRIMARY OUTCOMES:
The longitudinal trajectory of symptoms, endoscopy, and histology in pediatric EoE during routine clinical care | 10 years
  Outcome measures of symptoms, histology, endoscopy, and lab values such as peripheral eosinophilia and cortisol procured at each clinical and/or endoscopy visit will be entered and tracked in a UCSD/RCHSD de-identified database in order to understand their longitudinal trajectory during routine clinical care
The longitudinal trajectory of inflammatory markers in blood and biopsies in pediatric EoE during routine clinical care | 10 years
  The presence and severity of inflammatory markers and cells over time in specimens collected during routine endoscopy and biopsy will be measured to understand their alignment with outcome measures of symptoms, histology, and endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information and samples might be shared with other researchers at other institutions
Time Frame: Ongoing